CLINICAL TRIAL: NCT01520766
Title: Prefabricated Endodontic Posts: Glass Fiber Versus Titanium - A Randomized Controlled Pilot- Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Guido Sterzenbach, Principal Investigator, Dr. med. dent., Assistant Professor, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CC3-7.103
Record Dates: First submitted 2012-01-24; First posted 2012-01-30 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Endodontically Treated Teeth; Tooth Fractures
Keywords: glass fiber posts; titanium posts; postendodontic restoration; self-adhesive resin cement
MeSH Terms: conditions — Tooth, Nonvital; Tooth Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- glass fiber (Experimental)
  Interventions: Device: prefabricated glass fiber reinforced composite post
- titanium (Experimental)
  Interventions: Device: prefabricated titanium post

INTERVENTIONS:
Device: prefabricated titanium post — posts: diameter of 1.4 mm; length of 13 mm adhesively luted within the root canal using self-adhesive resin cement and direct composite cores using an etch-and-rinse adhesive were built up crown preparation was performed, while the finishing line for the final restoration was set at least 2 mm apical the composite build-up in dentin to ensure a proper dentin ferrule design
  Other Names: Fiberpoints Root Pins Titanium, Schuetz Dental Group
  Arms: titanium
Device: prefabricated glass fiber reinforced composite post — posts: diameter of 1.4 mm; length of 13 mm adhesively luted within the root canal using self-adhesive resin cement and direct composite cores using an etch-and-rinse adhesive were built up crown preparation was performed, while the finishing line for the final restoration was set at least 2 mm apical the composite build-up in dentin to ensure a proper dentin ferrule design
  Other Names: Fiberpoints Roots Pins Glass, Schuetz Dental Group
  Arms: glass fiber

SUMMARY:
A randomized parallel-group clinical pilot study was designed to evaluate the impact of glass fiber reinforced composite posts compared to prefabricated titanium posts on long term survival of adhesively restored endodontically treated abutment teeth.

DETAILED DESCRIPTION:
Compared to vital teeth the complication rate of restorations fixed on endodontically treated abutment teeth is higher. Endodontically treated teeth are more prone to fracture due to the higher amount of calcified tooth structure loss. To level the biological short coming the choice of the mechanically appropriate post material is still a major concern. There a two major approaches. One is to use a rigid material to stiffen the post-endodontic complex and the other is to use a material which shows dentin-like material properties to allow the post-endodontic complex to flex under load. It was aim of the presented randomised controlled trial to compare the survival rates of abutment teeth self-adhesively restored with either prefabricated glass-fiber reinforced composite posts or titanium posts.

The null-hypothesis was that there is no difference regarding survival rate between glass-fiber and titanium post restored endodontically treated abutment teeth with two or less remaining cavity walls.

ELIGIBILITY:
Inclusion Criteria:

* two or less cavity walls of the crown remaining,
* residual root canal thickness at the orifice of more than 1 mm,
* symptom free tooth with a root canal filling without radiologically visible periapical lesion,
* minimum of radiologic root-to-alveolar bone ratio of 2 after prospective crown lengthening,
* no or treated periodontitis with maximum probing depth of 4 mm and no bleeding on probing,
* tooth mobility not more than score II,
* willingness to return for follow-up examination for at least 5 years

Exclusion Criteria:

* tooth was aimed to serve as telescopic crown abutment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2003-01; Primary Completion 2004-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
loss of restoration for any reason | 84 months after post placement
  The patients were recalled at 3, 6, 12 month and thereafter in al yearly recall up to 84 month after post placement for clinical examination. The clinical examination was performed by one blinded dentist.

SECONDARY OUTCOMES:
tooth loss, post debonding, post fracture, vertical or horizontal root fracture, endodontic or periradicular conditions requiring endodontic re-treatment, secondary caries and failure of core build-up and loss of restoration due to technical failures | 84 month after post placement
  The clinical examination was performed by one blinded dentist. Follow-up examinations were performed with a dental probe to detect marginal gap formation of restorations. After 12 and 60 months radiographs were taken and examined by one operator (MN) to exclude the possibility of radiographic symptoms of failure, e.g. periodontal or periapical lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, CC3, Department of Prosthodontics, Geriatric Dentistry and Craniomandibular Disorders, Germany, Berlin, State of Berlin, Germany

REFERENCES:
- [Result] Naumann M, Sterzenbac G, Alexandra F, Dietrich T. Randomized controlled clinical pilot trial of titanium vs. glass fiber prefabricated posts: preliminary results after up to 3 years. Int J Prosthodont. 2007 Sep-Oct;20(5):499-503. PMID 17944340